CLINICAL TRIAL: NCT06590480
Title: An Expanded Access Program - Real-world Data Collection for VO in Combination With Nivolumab in Patients With Advanced Melanoma That Has Progressed on an Anti-PD-1 Containing Treatment Regimen
Brief Title: An Expanded Access Program for VO (RP1) in Combination With Nivolumab in Patients With Advanced Melanoma
Acronym: RPL-EAP-001
Status: No longer available | Type: Expanded Access
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RPL-EAP-001; RPL-EAP-001 (Other: Replimune Inc.)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Melanoma
Keywords: Advanced melanoma; Cutaneous melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: RP1 — Genetically modified Herpes Simplex Type 1 Virus
  Other Names: vusolimogene oderparepvec
Biological: Nivolumab — Anti-PD-1 Monoclonal Antibody
  Other Names: Opdivo

SUMMARY:
The purpose of this EAP is to provide expanded access (i.e., before marketing authorization) to vusolimogene oderparepvec (VO; herein referred to as VO) plus standard-of-care (SOC), nivolumab, for eligible patients diagnosed with advanced melanoma, who, in their treating physician's opinion, could benefit from this treatment.

DETAILED DESCRIPTION:
The objective of treating with VO is to directly reduce or eliminate tumors by lytic virus replication and to induce a systemic anti-tumor immune response leading to tumor immunity and durable clinical responses. Limited treatment options are available to those patients with advanced melanoma who have progressed while on an anti-PD-1 therapy regimen, and the duration of progression-free survival (PFS) is less than 6 months with overall survival (OS) being less than 3 years. The mechanism of VO complements that of anti-PD-1 therapy such that combining VO with an anti-PD-1 agent, such as nivolumab, will increase the number of tumor-reactive T cells (through the action of VO) and relieve CD8-T cell exhaustion (through the action of the anti-PD-1 therapy). Combining VO with nivolumab, is supported by evidence in syngeneic immune-competent murine models demonstrating an increased reduction in tumor volume compared with either VO or anti-PD-1 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the program:

1. Voluntary agreement to provide written informed consent and a willingness and ability to comply with protocol requirements.
2. Male or female ≥18 years old.
3. Histologically, cytologically, or clinically confirmed diagnosis of unresectable or metastatic Stage IIIb though IV/M1a through M1d cutaneous melanoma, as per AJCC staging system, 8th edition.
4. Prior treatment with an anti-PD-1-containing regimen as monotherapy or in combination (i.e., LAG-3).
5. Has ≥ 1 measurable and injectable lesion of ≥ 1 cm in longest diameter (or shortest diameter for lymph nodes).
6. Has adequate hematologic function including:

   1. White blood cell count ≥ 2.0 × 109/L
   2. Absolute neutrophil count ≥ 1.5 × 109/L
   3. Platelet count ≥ 75 × 109/L
   4. Hemoglobin ≥ 8 g/dL (without packed red blood cell transfusion within 2 weeks of dosing)
7. Has adequate hepatic function, including:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN; < 2.0 × ULN for patients with known Gilbert syndrome or liver metastases)
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN (≤ 5.0 × ULN, if liver metastases are present)
   3. Alkaline phosphatase (ALP) ≤ 2.5 × ULN (or ≤ 5.0 × ULN, if liver or bone metastases are present)
8. Has adequate renal function, defined as serum creatinine ≤ 1.5 × ULN or creatinine clearance ≤ 30.0 mL/minute/1.73 m2 (measured using Chronic Kidney Disease Epidemiology collaboration [CKD-EPI] formula)
9. Prothrombin time (PT) ≤ 1.5 × ULN (or international normalization ratio [INR] ≤ 1.3) and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Note: Patients which are on chronic anticoagulant therapy may be enrolled if the target international normalized ratio (INR) is ≤ 2.5. for patients requiring deep injection of VO, the INR must be < 1.5 at the time of injection.
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1.
11. Life expectancy of ≥ 3 months.
12. Male and female patients of reproductive potential must agree to avoid becoming pregnant or impregnating a partner and adhere to highly effective contraception requirement during treatment and for at 90 days after last dose of VO, or 5 months after last dose of nivolumab.
13. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test with a minimum sensitivity of 25 IU/L or equivalent units β-hCG within 7 days before the first dose of program treatment.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria will not be included in the program:

1. Eligibility for, or previous randomization in the Replimune clinical trial NCT06264180 (IGNYTE3 trial).
2. Prior treatment with anti-CTLA-4-directed therapy.
3. More than 2 lines of systemic therapy for advanced melanoma.
4. Known acute or chronic hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known acute or chronic hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected). Note: Patients who have been effectively treated are eligible for enrolment. Patients must be negative for HBsAg and HCV RNA.
5. Known human immunodeficiency virus (HIV) infection. Note: Testing for HIV is not required unless mandated by local health authority or clinically indicated.
6. Active significant herpetic infections or prior complications of herps simplex virus (HSV)-1 infection (e.g., herpetic keratitis or encephalitis) or requires intermittent or chronic use of systemic (oral or intravenous [IV]) antivirals with known antiherpetic activity (e.g., acyclovir). Note: Patients with sporadic cold sores may be enrolled as long as no active cold sores are present at the time of first dose of program treatment.
7. Had systemic infection requiring IV antibiotics or other serious active infection requiring antimicrobial, antiviral, or antifungal treatment within 14 days before dosing.
8. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis at time of screening. Patients with known CNS metastases are eligible if they have received SOC therapy for CNS disease (such as stereotactic radiosurgery or radical surgical resection followed by radiotherapy) and have disease stability on 2 subsequent scans performed at least at a 4-week interval.
9. Evidence of spinal cord compression or at high risk of spinal cord compression.
10. Serum lactate dehydrogenase > 2 × ULN.
11. Major surgery ≤ 2 weeks before starting program treatment.
12. No concurrent active malignancy requiring treatment.
13. History of significant cardiac disease including myocarditis or congestive heart failure (defined as New York Heart Association Functional Classification III or IV), or unstable angina, serious uncontrolled cardiac arrhythmia, cerebral vascular accident, or myocardial infarction within 6 months from first dose of VO.
14. History of life-threatening toxicity related to prior immune therapy except those that are unlikely to recur with standard countermeasures (e.g., hormone replacement after adrenal crisis).
15. History or evidence of psychiatric, substance abuse (including IV substance abuse) or any other clinically significant disorder, condition, or disease (with the exception of those described above) that, in the opinion of the treating physician would pose a risk to patient safety or interfere with the program evaluation, procedures, or completion.
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the program, interfere with the patient's participation for the full duration, or is not in the best interest of the patient to participate, in the opinion of the treating physician.
17. Active, known, or suspected autoimmune disease requiring systemic treatment.
18. History of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
19. Prior oncolytic virus therapy or other therapy given by intratumoral administration.
20. Was administered a live vaccine ≤ 28 days before the first dose of program treatment.
21. Systemic anticancer therapies within 5 half-lives or 4 weeks of the first dose, whichever is shorter.
22. Is currently participating in or has participated in a study of an investigational agent within 4 weeks before the first dose of program treatment.
23. Has received prior radiotherapy and has not recovered from radiotherapy.
24. Conditions requiring treatment with immunosuppressive doses (> 10 mg per day of prednisone or equivalent) of systemic corticosteroids other than for corticosteroid replacement therapy 14 days before enrollment. Note: Patients who require a brief course (≤ 7 days) or corticosteroids (e.g., as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded. Physiologic replacement doses of systemic corticosteroids are permitted, only if the dose does not exceed 10 mg/day prednisone equivalent.
25. History of allergy or sensitivity to program drug components (VO, nivolumab) or prior monoclonal antibody treatment.
26. Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks before treatment.
27. Patient is deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hash, MD, Study Director — Replimune Inc.